CLINICAL TRIAL: NCT00462358
Title: A Study of ARRY-520 in Patients With Advanced Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Array Biopharma, now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Sponsor
Organization: Array BioPharma (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ARRAY-520-101
Record Dates: First submitted 2007-04-18; First posted 2007-04-19 (Estimated); Last update posted 2020-09-28 (Actual); Status verified 2020-09

CONDITIONS: Advanced Solid Tumors
MeSH Terms: interventions — filanesib; Filgrastim; Granulocyte Colony-Stimulating Factor; Injections, Subcutaneous

ARMS (2):
- ARRY-520 (Experimental)
  Interventions: Drug: ARRY-520, KSP(Eg5) inhibitor; intravenous
- ARRY-520 + G-CSF support (Experimental)
  Interventions: Drug: ARRY-520, KSP(Eg5) inhibitor; intravenous; Drug: Filgrastim, granulocyte-colony stimulating factor (G-CSF); subcutaneous

INTERVENTIONS:
Drug: ARRY-520, KSP(Eg5) inhibitor; intravenous — Part 1: multiple dose, escalating; Part 2: multiple dose, single schedule.
Drug: Filgrastim, granulocyte-colony stimulating factor (G-CSF); subcutaneous — Part 1: standard of care; Part 2: standard of care.
  Arms: ARRY-520 + G-CSF support

SUMMARY:
This is a Phase 1 study during which patients with advanced solid tumors will receive investigational study drug ARRY-520.

This study has two parts. In the first part, patients with advanced solid tumors will receive increasing doses of study drug, with or without granulocyte-colony stimulating factor (G-CSF) support, in order to achieve the highest dose possible that will not cause unacceptable side effects. Approximately 15 patients (per schedule) from the US will be enrolled in Part 1 (Completed).

In the second part of the study, patients will receive the best dose of study drug determined from the first part of the study and will be followed to evaluate what side effects the study drug causes and what effectiveness it has, if any, in treating the cancer. Approximately 15 patients from the US will be enrolled in Part 2 (Completed).

ELIGIBILITY:
Key Inclusion Criteria:

* Histological or cytological evidence of malignancy.
* Advanced solid tumors that have recurred or progressed following standard therapy(ies).
* Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1 or 2.
* Adequate hematology counts and serum chemistry values.
* Additional criteria exist.

Key Exclusion Criteria:

* Treatment with an investigational product or device, or anti-neoplastic therapy (with the exclusion of hormone therapy where the therapy will continue at a standard dose throughout the study) within 28 days prior to the first dose of study drug.
* Major surgery within 28 days prior to the first dose of study drug.
* Radiotherapy (RT) within 28 days prior to the first dose of study drug (except if local RT to <5% of the bone marrow).
* Known positive serology for the human immunodeficiency virus (HIV), hepatitis C, and/or active hepatitis B.
* Additional criteria exist.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2007-04 (Actual); Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Establish the maximum tolerated dose (MTD) of study drug, with and without G-CSF. | Part 1
Characterize the safety profile of the study drug in terms of adverse events, clinical laboratory tests and electrocardiograms. | Part 1 and Part 2

SECONDARY OUTCOMES:
Characterize the pharmacokinetics of the study drug. | Part 1 and Part 2
Assess the efficacy of the study drug in terms of tumor response. | Part 1 and Part 2

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (2):
- United States (2):
  - Marlene and Stewart Greenebaum Cancer Center, Baltimore, Maryland
  - Wayne State University, Karmanos Cancer Institute, Detroit, Michigan